CLINICAL TRIAL: NCT01904396
Title: Identification of Carnitine-responsive Cardiomyopathy and Myopathy in Adult Patients With Dilated and/or Hypertrophic Cardiomyopathy and Limb Girdle Weakness.
Brief Title: Identification of Carnitine-Responsive Cardiomyopathy
Acronym: C001
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Hanna Faghfoury, Clinical and Metabolic Geneticist, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Carnitine001
Record Dates: First submitted 2013-07-15; First posted 2013-07-22 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Carnitine Deficiency
MeSH Terms: conditions — Systemic carnitine deficiency | interventions — Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CarnitineDeficient (Experimental): Patients identified with primary and secondary carnitine deficiency in the cardiomyopathy population will be prescribed with carnitine supplements to assess cardiac muscle function and status.
  Interventions: Drug: Carnitine

INTERVENTIONS:
Drug: Carnitine — Patients who are found to be carnitine deficient will be started on carnitine replacement and their heart function will be monitored on carnitine.
  Other Names: Carnitor

SUMMARY:
There are some adults with skeletal muscle weakness (called "myopathy") and heart muscle weakness (called "cardiomyopathy") who have low blood levels of a compound called carnitine as a cause of their problems. Carnitine is very important to energy production in muscles. In fact, there are reports of some people with carnitine deficiency who have developed myopathy and cardiomyopathy that was completely reversed with carnitine treatment. The main objective of our project is to determine the number of patients who have carnitine deficiency as a cause of their myopathy and cardiomyopathy. The investigators will be measuring carnitine levels in 1000 patients with cardiomyopathy and will describe the specific features in all the study patients to see if there are any trends that may help us predict which patients with muscle weakness are at risk of developing low carnitine levels. The investigators will be treating patients with low carnitine levels with carnitine and observing them to see if their cardiomyopathy and their muscle weakness improve. Knowing the exact percentage of myopathy and cardiomyopathy patients with carnitine deficiency may allow for screening of patients in a cheap and targeted way to treat the serious complication of this condition, including heart failure and sudden death.

DETAILED DESCRIPTION:
The primary objective of this research is to determine the prevalence of primary and secondary (genetic and acquired) carnitine deficiency in patients with limb girdle weakness and hypertrophic or idiopathic dilated cardiomyopathy where an underlying cause is unknown. Identification and treatment with carnitine may potentially reverse or halt heart failure and skeletal muscle weakness in these patients.

Specific aims:

1. To ascertain the prevalence of primary and secondary carnitine deficiency in a population of adults with myopathy and hypertrophic and dilated cardiomyopathy of unknown etiology
2. To describe the demographic and phenotypic characteristics of patients with myopathy and dilated or hypertrophic cardiomyopathy who have primary and secondary carnitine deficiency
3. To measure the motor and cardiovascular response to carnitine supplementation in patients with myopathy, cardiomyopathy and carnitine deficiency

ELIGIBILITY:
Inclusion Criteria:

* An adult patient (>18 years) with a diagnosis of either hypertrophic or dilated cardiomyopathy, for which the underlying etiology of the cardiomyopathy is unknown.

Exclusion Criteria:

* A history of ischemia
* A documented or suspected infection including HIV
* A history of severe longstanding hypertension
* A history of valvular heart disease
* A history of chemotherapy exposure
* A history of alcohol abuse
* Carnitine supplementation at the time of recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Serum Carnitine Concentration | Baseline
  Measurement of free and total serum carnitine concentrations will be performed using isotope-dilution mass spectrometry.

SECONDARY OUTCOMES:
Echocardiographic Measures | Baseline, every 6m for up to 2 years
  Measurements include:
  Septal diameter Left Ventricular (LV) mass LV ejection fraction LV end-systolic volume LV end-diastolic measure
B-Natriuretic Peptide (BNP) | Baseline, every 6m for up to 2 years
  An elevated BNP level is a marker of increased LV filling pressures and LV dysfunction and is highly correlated with severity of, and prognosis in, heart failure. BNP testing is routinely performed at the cardiac clinic at University Health Network to determine treatment response and to assist with risk stratification prognostication in patients with heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Faghfoury Hannaneh, MD, Principal Investigator — University Health Network, Toronto, Ontario; Ingrid Tein, MD, Principal Investigator — The Hospital for Sick Children, Toronto, Ontario
Locations (1):
- University Health Network, Toronto, Ontario, Canada